CLINICAL TRIAL: NCT01001260
Title: Biosynthesis of PGD2 in Vascular Injury
Brief Title: PGD2 Formation in Vascular Injury
Acronym: PGD2
Status: Terminated | Type: Observational
Why Stopped: Unable to find subjects that met inclusion/exclusion criteria.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 804975; American Heart Association
Record Dates: First submitted 2009-10-14; First posted 2009-10-26 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Stable Angina
Keywords: Prostaglandins; vascular injury
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Angina, Stable; Vascular System Injuries | interventions — nitroxy-butyl-acetylsalicylic acid; Aspirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * Specimens:
    3 urine collections will be obtained (Prior to PTCA, During PTCA and Post PTCA)
  * Genetic Testing:
  analysis of the association of SNPs in Cox genes with variability in selectively or in the PGEs genes in quantitative biosynthesis of PGD2 and related compounds.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No Aspirin Treatment
  Interventions: Drug: No ASA
- 81 mg Aspirin Treatment
  Interventions: Drug: Low dose ASA
- 325 mg Aspirin
  Interventions: Drug: 325 mg ASA

INTERVENTIONS:
Drug: No ASA — Alternative antiplatelet therapy instead of aspirin
  Groups: No Aspirin Treatment
Drug: Low dose ASA — Low dose aspirin (81mg) prior to PTCA
  Groups: 81 mg Aspirin Treatment
Drug: 325 mg ASA — high dose of aspirin prior to PTCA
  Groups: 325 mg Aspirin

SUMMARY:
To investigate the biosynthesis of PGD2 during percutaneous transluminal coronary angioplasty (PTCA) procedure.

DETAILED DESCRIPTION:
A) To determine whether biosynthesis of PGD2 is altered in response to vascular injury in humans

B) Patients will be grouped base on their aspirin using status. Three groups of no aspirin but an alternative anti-platelet medicine, low dose (81 mg) aspirin, high dose 325 mg aspirin will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with existing CAD admitted for elective PTCA:

  1. Treated with any dose of aspirin daily for at least 5 days, with special interest in those treated with 81 mg aspirin daily or
  2. Treated with an alternative antiplatelet therapy, such as clopidogrel, due to aspirin hypersensitivity or PMDs preference or
  3. No aspirin therapy at all
* Patients presenting to the ER with Acute Coronary Syndrome(ACS)who will have a PTCA
* Patients with stable angina or positive stress tests scheduled for a cardiac catheterization

Exclusion Criteria:

* History of unstable diabetes (hgb A1c>8 or FBS> 200)
* Uncontrolled hypertension (SBP > 180, DBP >100)
* History of an acute confounding disease as judged on clinical screen that according to the investigator may interfere with interpretation of the study results, or compromise the safety of a potential subject.
* Patients who have taken NSAIDS or COX-2 inhibitors other than aspirin, for at least 10 days prior to PTCA

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to have PTCA
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2007-08; Primary Completion 2011-02 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The increment of PGD2 synthesis reflected by an novel biomarker of urinary PGD2 metabolite. | 18-48 hours - which includes 24 hours before the procedure through 18 hours after the procedure for a continuous urine collection.

SECONDARY OUTCOMES:
Whether aspirin could blunt the increment of PGD2 if there is. | 18-48 hours - which includes 24 hours before the procedure through 18 hours after the procedure for a continuous urine collection.

CONTACTS AND LOCATIONS:
Overall Officials: Garret FitzGerald, MD, Principal Investigator — University of Pennsylvania; Wenliang Song, MD, Principal Investigator — University of Pennsylvania